CLINICAL TRIAL: NCT03263767
Title: Phase II Study Testing Prophylaxis Feasibility of Graft Versus Host Disease With Only High Dose Cyclophosphamide Post-transplantation for Patients Eligible to a Reduced-intensity Conditioning Regiment Prior to Allogenic Transplantation With a Compatible Familial or Non-familial Donor.
Brief Title: Post Transplant Cyclophosphamide (PTCY) as Sole Graft Versus Host Disease (GVHD) Prophylaxis for Matched Allotransplant: CYRIC
Acronym: CYRIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Security criteria (MTD)
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0435
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Graft Versus Host Disease
Keywords: Peripheral haemopoietic stem cell transplant; High dose cyclophosphamide; acute GVHD; allogenic transplantation; RIC (reduced-intensity conditioning)
MeSH Terms: conditions — Graft vs Host Disease | interventions — fludarabine; Clofarabine; Cyclophosphamide; Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LYMPHOID HEMOPATHY without ATG (Experimental): patients with lymphoid hemopathy
  Interventions: Drug: Fludarabine; Radiation: Full body irradiation; Drug: Cyclophosphamide; Other: stem cell transplantation; Other: nuclear cells
- MYELOID HEMOPATHY without ATG (Experimental): patients with myeloid hemopathy
  Interventions: Drug: Clofarabine; Radiation: Full body irradiation; Drug: Cyclophosphamide; Other: stem cell transplantation; Other: nuclear cells
- LYMPHOID HEMOPATHY witH ATG (Experimental): patients inclued after 14 dec 2020, received a conditionnement regimen with ATG on Day -2 to reduce GVHD GRADE 1-2 incidence
  Interventions: Drug: Fludarabine; Radiation: Full body irradiation; Drug: Cyclophosphamide; Other: stem cell transplantation; Other: nuclear cells; Drug: Thymoglobulin Injectable Product
- MYELOID HEMOPATHY with ATG (Experimental): patients inclued after 14 dec 2020, received a conditionnement regimen with ATG on Day -2 to reduce GVHD GRADE 1-2 incidence
  Interventions: Drug: Clofarabine; Radiation: Full body irradiation; Drug: Cyclophosphamide; Other: stem cell transplantation; Other: nuclear cells; Drug: Thymoglobulin Injectable Product

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m² Intravenous 5 days from Day-6 to Day-2
  Arms: LYMPHOID HEMOPATHY witH ATG; LYMPHOID HEMOPATHY without ATG
Drug: Clofarabine — 30 mg/m² Intravenous 5 days from Day-6 to Day-2
  Arms: MYELOID HEMOPATHY with ATG; MYELOID HEMOPATHY without ATG
Radiation: Full body irradiation — 2 grays at Day-1
Drug: Cyclophosphamide — 14 mg/kg intravenous 2 days at Day - 6 and day -5
Drug: Cyclophosphamide — 50 mg/kg intravenous 2 days at day +3 and day +4
  Other Names: hight dose
Other: stem cell transplantation — at D0 intraveinous Depending on donor : the stem cells will be extracted from blood (CD34+) or from bone marrow (CD34+ and nuclear cells)
  Other Names: graft
Other: nuclear cells — CD3+ cells if needed after transplantation
  Other Names: Donor Lymphocytes Injection (DLI)
Drug: Thymoglobulin Injectable Product — At day -2 2.5 mg/kg for patients inclued after 14 dec 2020
  Other Names: ATG
  Arms: LYMPHOID HEMOPATHY witH ATG; MYELOID HEMOPATHY with ATG

SUMMARY:
Acute or chronic graft versus host disease is still the major complication of stem cells transplantation regarding morbidity and mortality.

Recently, high dose cyclophosphamide utilization early after post-transplantation (day+ 3 and +4) not only for patients with HLA- haploidentical donor but also for patients with Human Leukocyte Antigen (HLA)-compatible donor, showed a great control of graft versus host disease after transplantation, allowing to consider stopping immunosuppressive treatment after the transplantation (Neoral=cyclosporine, cell-cept=mycophenolate mofetil). Indeed, this step has already been completed in myeloablative transplantation in adult patients.

This approach could enable to avoid in the end several complications related to long term immunosuppressive drugs administration, while promoting quicker immunity recovery.

DETAILED DESCRIPTION:
The BALTIMORE conditioning regiment will be used in this study with peripheral stem cell transplantation and fludarabine will be replaced by clofarabine for myeloid diseases (Acute Myeloide Leukemia, Myelodysplasia , myelofibrosis, Chronic Myeoloid Leukemia..) because of better antitumoral activity in this setting.

ELIGIBILITY:
Inclusion Criteria:

* adults ≤ 70 years old
* indication to stem cells transplantation with reduced-intensity conditioning regimen
* with a HLA-compatible familial 10/10 or non-familial donor
* Written signed informed consent form
* woman with childbearing potential under efficient control birth method during the trial and up to 12 months after cyclophosphamide stop
* men under efficient control birth method during the trial and up to 6 months after cyclophosphamide stop
* Negative serology to B and C hepatitis and to HIV
* Affiliated to social security

Exclusion Criteria:

* - Eligible to myeloablative contioning regimen
* Other progressive malignancy disease or history of prior other malignancy in the last two years, with the exception of: curatively treated basal cell carcinoma or carcinoma in situ of the cervix
* Progressive mental illness disease
* Pregnant or Breastfeeding woman
* woman with childbearing potential without any efficient control birth
* Serious concomitant infection and not controlled
* Contra-indications to allogenic transplantation, especially:

  * Cardiac: left ventricular ejection fraction <45% assessed by transthoracic echography or isotopic method (isotopic gamma-angiography)
  * Respiratory: DLCO limiting fludarabine and busulfan use (DLCO< 40% of theorical value)
  * Renal: creatinine clearance < 60ml/min (MDRD method)
  * Hepatic: transaminases >5 Uper Per Normal (UPN) or bilirubin> 2 UPN
* Contra-indications to cyclophosphamide:

  * Urinary tract infections
  * Acute urothelial toxicity due to cytotoxic chemotherapy or to radiotherapy
  * Obstruction of urines flow
  * Pre-existing hemorrhagic cystitis
  * Yellow fever vaccination
* Cardiac condition preventing high dose cyclophosphamide utilization :

  * New York Heart Association (NYHA) functional class II, III or IV
  * Rhythmic, valvular or ischemic cardiomyopathy
* Minor
* Patient under guardianship or curatorship
* Patient under judicial protection
* Known or suspected hypersensitivity to cyclophosphamide
* Known or suspected hypersensitivity to rabbit proteins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 and 4 acute GVHD cortico-resistant | 100 days after transplantation
  acute GVHD will be evaluated from International Mount Sinai criteria

SECONDARY OUTCOMES:
Engraftment | one year
  number of days in aplasia (neutrophils< 0.5 Giga/L and platelets<20 G/l, number of transfusions (red blood and platelets)
Engraftment | one year
  chimerism
disease free survival (DFS) | one year, the last follow-up visit
  blood and bone marrow analysis
Overall survival (OS) | one year, the last follow-up visit
  clinical follow-up
graft and relapse free survival | one year
  time between Day O and relapse
chronic GVHD | one year
  chronic GVHD will be assessed with NCI criteria for evaluation of chronic GVHD
non relapse mortality (NRM) | last follow-up visit
  number of death unrelated to relapse or disease progression
Chimerism | 1, 2, 3, 6 and 12 months after transplantation
  proportion of full and mixed donor chimerism
Immune reconstitution | 3, 6 and 12 months after transplantation
  lymphocytes, monocytes, T4, T8, Natural Killer (NK), B cells rates
Identification of ghost factors associated with GVHD | one year
  Statistical Models to Identify Subjects with Ghost Prognosis Factors Nguyen JM. 2015
Adverse events of grade 3 and 4 after transplantation | one year
  time of occurring and frequency of grade 3 and grade 4 adverse events (CTCAE criteria)
Infections frequency | one year
  time of occurring and frequency of viral (CytoMegalo Virus, Epstein Barr virus , BKV, adenovirus), bacterial, parasite and yeast infections, evaluated by Polymerase Chain Reaction (PCR), blood and urines cultures, biopsy if applicable
compare OS between patients with ATG and patients without ATG | one year, last follow-up visit
  OS
compare grade 2-4 and 3-4 acute GVHD between patients with ATG and patients without ATG | one year
  acute GVHD will be evaluated from International Mount Sinai criteria
compare chronic GVHD between patients with ATG and patients without ATG | one year
  chronic GVHD will be assessed with NCI criteria for evaluation of chronic GVHD
compare DFS between patients with ATG and patients without ATG | one year, last follow-up visit
  DFS
compare Relapse between patients with ATG and patients without ATG | one year, last follow-up visit
  Relapse
compare NRM between patients with ATG and patients without ATG | one year, last follow-up visit
  NRM
compare Infections frequency between patients with ATG and patients without ATG | one year
  time of occurring and frequency of viral (CytoMegalo Virus, Epstein Barr virus , BKV, adenovirus), bacterial, parasite and yeast infections, evaluated by Polymerase Chain Reaction (PCR), blood and urines cultures, biopsy if applicable

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Uh, Nantes, France

IPD SHARING:
Plan to Share IPD: No